CLINICAL TRIAL: NCT00530920
Title: A Multicenter, Randomized, Open Label, Clinical Trial to Evaluate Three Doses of Tipranavir Boosted With Ritonavir (500 mg/200 mg qd, 250 mg/100 mg Bid and 500 mg/100 mg Bid) by Assessing the Steady-state Pharmacokinetics and Short-term Efficacy and Safety in HIV-1 Positive Treatment naïve Patients
Brief Title: Tipranavir/Ritonavir Low Dose Pharmacokinetics in Treatment Naive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1182.107
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

INTERVENTIONS:
Drug: tipranavir
Drug: ritonavir

SUMMARY:
The purpose of this study is to identify an optimal dose combination(s) of tipranavir (TPV) and ritonavir (RTV) for antiretroviral treatment naïve HIV-1 infected patients that can be used in pivotal trial by assessing the steady-state pharmacokinetics and short-term efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in accordance with GCP and local regulatory requirements prior to trial participation.
* HIV-1 infected men and non-pregnant women who are treatment naïve, with positive serology (EIA) confirmed by Western blot.
* Age > 18 and < 65 years.
* CD4 > 200 cells/mm3
* Viral load (HIV-1 mRNA viral load) > 5,000 copies/mL.
* Ability to swallow multiple large capsules without difficulty.
* Acceptable laboratory values that indicate adequate baseline organ function at screening visit.
* Laboratory values are considered to be acceptable if the severity of any parameter is = < Grade 2, based on the DAIDS/ACTG Grading Scale (see Appendix 10.2).
* Acceptable medical history, physical examination, and 12-lead ECG at screening
* Willingness to abstain from the following starting 2 weeks prior to administration of any study medication and up until the end of the study:

  o Grapefruit or grapefruit juice, Seville oranges, St. John's Wort, and Milk Thistle.
* Willingness to abstain from alcohol 3 days prior to administration of any study medication up to the end of the study.
* Willingness to abstain from the following starting 3 days prior to PK sampling:

  o Garlic supplements and methylxanthine containing foods or drinks (including coffee, tea, cola, energy drinks, chocolate, etc.).
* Willingness to abstain from over-the-counter herbal medications for the duration of the study.
* Willingness to abstain from any over the counter medication 7 days prior to administration of any study medication (including vitamins, minerals, dietary supplements and antacids) during the study until completion of the post study assessments.

Exclusion Criteria:

* Female patients of reproductive potential who:

  * Have positive serum pregnancy test.
  * Have not been using a barrier method of contraception for at least 3 months prior to participation in the study.
  * Are not willing to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and 60 days after completion/termination of the trial.
  * Are breast-feeding.
* Suspected or documented seroconversion within last 6 months
* Participation in another trial with an investigational medicine within 2 months prior to Day 0 of this study.
* Use of any pharmacological contraceptive (including oral, patch or injectable contraceptives) within 1 month prior to Day 0 and for the duration of the study.
* Use of hormone replacement therapy within 1 month prior to Day 0 and anytime during the study.
* History of acute illness within 30 days prior to Day 0.
* Have evidence of active or acute HBV or HCV.
* Alcohol or substance abuse within 1 year prior to screening or during the study.
* Patients with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering TPV.
* Patients who have taken (within 7 days prior to Day 0) any over-the-counter or prescription medication that, in the opinion of the investigator in consultation with the BI clinical monitor, might interfere with absorption, distribution, or metabolism of the study medications.
* Known hypersensitivity to any ingredients of the test drug.
* Inability to adhere to the protocol.
* Genotypic resistance to tipranavir (defined as a TPV mutation score > 4).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- Germany (4):
  - 1182.107.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1182.107.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 1182.107.49003 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1182.107.49001 Boehringer Ingelheim Investigational Site, München
- Italy (4):
  - 1182.107.39001 Boehringer Ingelheim Investigational Site, Antella (fi)
  - 1182.107.39009 Boehringer Ingelheim Investigational Site, Bari
  - 1182.107.39007 Boehringer Ingelheim Investigational Site, Ferrara
  - 1182.107.39011 Boehringer Ingelheim Investigational Site, Palermo
- Spain (4):
  - 1182.107.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.107.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.107.34003 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1182.107.34004 Boehringer Ingelheim Investigational Site, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily: Tipranavir 500 mg boosted with ritonavir 200 mg given once daily
- Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily: Tipranavir 250 mg boosted with ritonavir 100 mg given once daily
- Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily: Tipranavir 500 mg boosted with ritonavir 100 mg given twice daily
Period: Overall Study
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Started | 30 | 27 | 28
Completed | 30 | 25 | 24
Not Completed | 0 | 2 | 4
Not completed — Randomized but not treated | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set, includes all patients that were randomized and were documented to have received at least one dose of investigational treatment
Groups:
- Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily: Tipranavir 250 mg boosted with ritonavir 100 mg given twice daily
- Total: Total of all reporting groups
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily | Total
Number analyzed (Participants) | 30 | 25 | 28 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (7.54) | 36.9 (8.04) | 36.4 (8) | 35.3 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 7
  Male | 28 | 24 | 24 | 76

OUTCOME MEASURES:

1. Primary Outcome: Viral Load (log10 Copies/mL) Change From Baseline (Last Observation Carried Forward (LOCF))
Time Frame: Baseline (Day 0) to Final (Day 14)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Log10 copies/mL
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 28
Log10 copies/mL | -1.43 [-1.66 to -1.24] | -1.55 [-1.70 to -1.37] | -1.47 [-1.66 to -1.09]
Statistical Analysis 1: Comparison: Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily; NULL HYPOTHESIS (H0): Median viral load reduction from baseline >1.2 log10 copies/mL within each group; Test type: Superiority or Other; p = 0.997, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.43
Statistical Analysis 2: Comparison: Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily; NULL HYPOTHESIS (H0): Median viral load reduction from baseline >1.2 log10 copies/mL within each group; Test type: Superiority or Other; p = 1, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.55
Statistical Analysis 3: Comparison: Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily; NULL HYPOTHESIS (H0): Median viral load reduction from baseline >1.2 log10 copies/mL within each group; Test type: Superiority or Other; p = 0.998, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.47

2. Secondary Outcome: Apparent Oral Clearance I(Cl/F) of Tipranavir
Description: Tipranavir pharmacokinetics - Clearance (CL) is defined as the dose of a drug divided by the area-under-the-concentration-time curve (AUC), ie. CL = Dose / AUC. For extravascu-lar models the fraction of dose absorbed cannot be estimated, therefore "clear-ance" for these models is actually Cl/F where F is the fraction of the drug dose which is absorbed.
Time Frame: Final (Day 14)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
L/h | 1.45 (26.79) | 1.43 (26.77) | 1.57 (35.40)

3. Secondary Outcome: Area Under the Curve(AUC) of Tipranavir 24 h for Once Daily (QD) and AUC 12 h for Twice Daily (BID)
Description: Tipranavir (TPV) pharmacokinetics
Time Frame: Final (Day 13 for QD, Day 14 for BID)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*uM
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 29 | 25 | 22
h*uM | 571.3 (27.3) | 289.3 (26.8) | 538.2 (36.4)

4. Secondary Outcome: Concentration-24 Hour (hr) Post Dose of Tipranavir - (Cp 24 h for QD and 12 hr Post Dose (CP 12h) for BID
Description: TPV pharmacokinetics
Time Frame: Final (Day 13 for QD, Day 14 for BID)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: uM
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 29 | 25 | 22
uM | 3.26 (92.4) | 10.27 (49.4) | 17.75 (71.7)

5. Secondary Outcome: Trough Concentration (Cmin) of Tipranavir
Description: TPV pharmacokinetics
Time Frame: Final (Day 13 for QD, Day 14 for BID)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: uM
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 29 | 25 | 22
uM | 2.8 (106.8) | 12.73 (53.1) | 21.26 (86.8)

6. Secondary Outcome: Maximum Concentration (Cmax) of Tipranavir
Description: TPV pharmacokinetics
Time Frame: Final (Day 13 for QD, Day 14 for BID)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: uM
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 29 | 25 | 22
uM | 54.64 (20.2) | 36.98 (19.9) | 69.66 (26.5)

7. Secondary Outcome: Volume of Distribution (V/F) of Tipranavir
Description: Tipranavir pharmacokinetics
Time Frame: Final (Day 14)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
L | 10.02 (14.33) | 9.33 (9.17) | 9.39 (12.34)

8. Secondary Outcome: Terminal Half-Life (t1/2) of Tipranavir
Description: Tipranavir pharmacokinetics
Time Frame: Final (Day 14)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
h | 4.79 (26.3) | 4.51 (22.4) | 4.14 (33.6)

9. Secondary Outcome: Time to Cmax (Tmax) of Tipranavir
Description: Tipranavir pharmacokinetics
Time Frame: Final (Day 14)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
h | 3.07 (14.7) | 2.34 (15.2) | 2.38 (16.6)

10. Secondary Outcome: AUC 24 of Ritonavir for QD and AUC 12 of Ritonavir for BID
Description: Ritonavir pharmacokinetics
Time Frame: Final (Day 13 for QD, Day 14 for BID)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*uM
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
h*uM | 5.05 (44.0) | 2.25 (47.0) | 1.74 (48.9)

11. Secondary Outcome: Cp 24 h of Ritonavir for QD and CP 12 h of Ritonavir for BID
Description: Ritonavir pharmacokinetics
Time Frame: Final (Day 13 for QD, Day 14 for BID)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: uM
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
uM | 0.005 (206.2) | 0.039 (134.0) | 0.025 (129.9)

12. Secondary Outcome: Apparent Oral Clearance I(Cl/F) of Ritonavir
Description: Ritonavir pharmacokinetics
Time Frame: Final (Day 13 for QD, Day 14 for BID)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
L/h | 39.6 (44.0) | 44.4 (47.0) | 57.4 (48.9)

13. Secondary Outcome: Volume of Distribution (V/F) of Ritonavir
Description: Ritonavir pharmacokinetics
Time Frame: Final (Day 14)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
L | 97.5 (26.8) | 90.8 (24.7) | 88.9 (28.7)

14. Secondary Outcome: Terminal Half-Life (t1/2) of Ritonavir
Description: Ritonavir pharmacokinetics
Time Frame: Final (Day 14)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
Hours | 1.71 (45.5) | 1.42 (59.5) | 1.07 (56.1)

15. Secondary Outcome: Tmax of Ritonavir
Description: Ritonavir pharmacokinetics
Time Frame: Final (Day 14)
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
h | 2.84 (23.9) | 2.33 (24.9) | 2.05 (28.8)

16. Secondary Outcome: Cmax of Ritonavir
Description: Ritonavir pharmacokinetics
Time Frame: Visits baseline, 5, 7, 9 and 13 or 14
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: uM
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
uM | 0.632 (32.5) | 0.346 (30.7) | 0.291 (34.7)

17. Secondary Outcome: Clinical Abnormal Findings in Laboratory and Physical Examination
Time Frame: Screening through the end of the study (14 days)
Population: Treated set.
Measure: Number; unit: participants
Groups:
- Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily: Tipranavir 500 mg boosted with ritonavir 200 mg given once daily
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Number analyzed (Participants) | 30 | 25 | 24
participants
  Alanine aminotransferase (ALT) increased | 0 | 0 | 1
  Aspartate aminotransferase (AST) increased | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 14 days, from first treatment until last treatment
Arm/Group | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/25 | 1/28
Other Adverse Events (participants affected / at risk) | 17/30 | 9/25 | 15/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily (N=30) | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily (N=25) | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily (N=28)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increaset (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tipranavir With Ritonavir (TPV/r) 500/200 mg Once Daily (N=30) | Tipranavir With Ritonavir (TPV/r) 250/100 mg Twice Daily (N=25) | Tipranavir With Ritonavir (TPV/r) 500/100 mg Twice Daily (N=28)
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 3 | 11
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 4
Fatigue (General disorders) | 1 | 3 | 2
Dizziness (Nervous system disorders) | 2 | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 4
Insomnia (Psychiatric disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.